CLINICAL TRIAL: NCT01297725
Title: Sharp Versus Blunt Fascial Incision at Caesarean Section: A Prospective Randomized Double-blinded Case-Control Study With the Case as it's Own Control.
Brief Title: Sharp Versus Blunt Fascial Incision at Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Anna Aabakke, Anna Aabakke, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Fascia Study; H-2-2010129 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Cesarean section[*methods]; Fascia [*surgery]; Randomized Controlled Trial; Abdominal Wall [*surgery]; Pain, postoperative; Surgical wound infection
MeSH Terms: conditions — Pain, Postoperative; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right sharp, left blunt (Experimental): Blunt fascial entry on the left side of the midline and sharp fascial entry on the right side of the midline.
  Interventions: Procedure: Blunt left, sharp right
- Right blunt, left sharp (Experimental): Blunt fascial entry on the right side of the midline and sharp fascial entry on the left side of the midline.
  Interventions: Procedure: Blunt right, sharp left

INTERVENTIONS:
Procedure: Blunt right, sharp left — Blunt fascial entry on the right side of the midline and sharp fascial entry on the left side of the midline.
  Arms: Right blunt, left sharp
Procedure: Blunt left, sharp right — Blunt fascial entry on the left side of the midline and sharp fascial entry on the right side of the midline.
  Arms: Right sharp, left blunt

SUMMARY:
The purpose of this study is to compare sharp and blunt fascial entry during caesarean section on the same patient. The study is performed on woman having cesarean section for the first time and who have not previously had lower abdominal surgery done. The following parameters are registered:

1. The preferred side evaluated by the patient 3 months postoperatively.
2. The patient evaluated difference in pain on the right vs. left side 1, 3 and 7 days and 1 and 3 months postoperatively.
3. The rate and side of infection.

ELIGIBILITY:
Inclusion Criteria:

* Woman having caesarean section for the first time
* Woman, who have had no previous lower abdominal surgery
* Woman who speak and understand Danish
* Woman who can give informed consent

Exclusion Criteria:

* Diabetes Mellitus (This does not include gestational diabetes)
* Infection
* Regular treatment with immunosuppressives
* Alcohol or drug abuse
* Age under 18 years old
* Chronic pain disease eg. fibromyalgia, rheumatoid arthritis
* BMI over 35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Preferred side of the scar evaluated by the patient 3 months postoperatively | 3 months
  The overall preference of scar side - left, right or no difference - taking the entire postoperative 3 months into account as evaluated by the patient.

SECONDARY OUTCOMES:
The difference in pain between the two sides of the scar | 1, 3 and 7 days postoperatively
  Difference in painscore between the two ends of the scar on the 1st, 2nd and 7th postoperative day. Pain is registered by a score on a vas-scale from 0-10.
The difference in pain between the two sides of the scar | 1 and 3 months postoperatively
  Description: Difference in painscore between the two ends of the scar one and three months postoperatively. Pain is registered by a score on a vas-scale from 0-10.
Pain on the two sides of the scar | 1, 3 and 7 days postoperatively
  Pain in the two ends of the scar registered by a score on a vas-scale from 0-10 1, 3 and 7 days postoperatively.
Pain in the two sides of the scar | 1 and 3 months postoperatively
  Pain in the two sides of the scar is registered by a score on a vas-scale from 0-10 1 and 3 months postoperatively.
Infection | 7 days
  The rate of postoperative infection and what side of the scar - right or left -that is infected.
Infection | 1 and 3 months postoperatively
  The rate of postoperative infection and what side of the scar - right or left -that is infected.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jørgen Secher, Professor, M.D., Study Chair — Dep. Gynaecology and Obstetrics, Hvidovre University Hospital; Anna Aabakke, M.D., Principal Investigator — Dep. Gynaecology and Obstetrics, Holbaek Hospital
Locations (2):
- Denmark (2):
  - Department of Gynaechology and Obstetrics, Holbaek Hospital, Holbæk
  - Department of Gynaecology and obstetrics, Hvidovre University Hospital, Hvidovre

REFERENCES:
- [Background] Nikolajsen L, Sorensen HC, Jensen TS, Kehlet H. Chronic pain following Caesarean section. Acta Anaesthesiol Scand. 2004 Jan;48(1):111-6. doi: 10.1111/j.1399-6576.2004.00271.x. PMID 14674981
- [Background] Jenkins TR. It's time to challenge surgical dogma with evidence-based data. Am J Obstet Gynecol. 2003 Aug;189(2):423-7. doi: 10.1067/s0002-9378(03)00587-8. PMID 14520211
- [Background] CAESAR study collaborative group. Caesarean section surgical techniques: a randomised factorial trial (CAESAR). BJOG. 2010 Oct;117(11):1366-76. doi: 10.1111/j.1471-0528.2010.02686.x. PMID 20840692
- [Background] CORONIS Trial Collaborative Group. The CORONIS Trial. International study of caesarean section surgical techniques: a randomised fractional, factorial trial. BMC Pregnancy Childbirth. 2007 Oct 22;7:24. doi: 10.1186/1471-2393-7-24. PMID 18336721
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Background] Mathai M, Hofmeyr GJ. Abdominal surgical incisions for caesarean section. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD004453. doi: 10.1002/14651858.CD004453.pub2. PMID 17253508
- [Background] Franchi M, Ghezzi F, Raio L, Di Naro E, Miglierina M, Agosti M, Bolis P. Joel-Cohen or Pfannenstiel incision at cesarean delivery: does it make a difference? Acta Obstet Gynecol Scand. 2002 Nov;81(11):1040-6. doi: 10.1034/j.1600-0412.2002.811108.x. PMID 12421172
- [Background] Holmgren G, Sjoholm L, Stark M. The Misgav Ladach method for cesarean section: method description. Acta Obstet Gynecol Scand. 1999 Aug;78(7):615-21. PMID 10422908
- [Background] Stark M, Finkel AR. Comparison between the Joel-Cohen and Pfannenstiel incisions in cesarean section. Eur J Obstet Gynecol Reprod Biol. 1994 Feb;53(2):121-2. doi: 10.1016/0028-2243(94)90218-6. PMID 8194647
- [Background] Mathai M, Ambersheth S, George A. Comparison of two transverse abdominal incisions for cesarean delivery. Int J Gynaecol Obstet. 2002 Jul;78(1):47-9. doi: 10.1016/s0020-7292(02)00061-9. No abstract available. PMID 12113971
- [Background] Bolla D, Schöning A, Drack G, Hornung R. Technical aspects of the cesarean section. Gynecol Surg 2010;7:127-32.
- [Derived] Aabakke AJ, Hare KJ, Krebs L, Secher NJ. Sharp compared with blunt fascial incision at cesarean delivery: a randomized controlled trial with each case as her own control. Eur J Obstet Gynecol Reprod Biol. 2014 Jan;172:40-5. doi: 10.1016/j.ejogrb.2013.10.029. Epub 2013 Nov 5. PMID 24275233